CLINICAL TRIAL: NCT05571228
Title: Be Outspoken and Overcome Stigmatizing Thoughts (BOOST) Group for Early Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Professor and Director of Clinical Training Department with the Psychology, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYC-242-20
Record Dates: First submitted 2022-01-17; First posted 2022-10-07 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Psychosis
Keywords: Early Psychosis; Remote treatment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Consultation with our lived-experience advisory group, consisting of service-users and family members, supports our decision to use a single-arm, non-randomized trial design. All participants recruited into the study will receive the intervention. Results of single arm interventions can provide rich data using data analytic techniques such as Reliable Change Index and will allow us to examine mediators of change from the intervention to continue to refine its efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internalized stigma group (Experimental): BOOST is an 8 session group intervention, delivered over 4 weeks. The program uses evidence based therapeutic techniques and integrates cognitive behavioural therapy and peer support to reduce or prevent the internalization of stigma in early psychosis. Sessions 1-4 focus on dispelling stigmatizing myths about psychosis and evaluating the accuracy of group members or societies stigmatizing beliefs in order to normalize experiences associated with and reactions to the symptoms of psychosis. Sessions 5-8 teach behavioural approaches for self-empowerment through social skills training, development of assertiveness skills, and goal setting. Role-plays that are specific to young people with psychosis, which were co-developed with people with lived experience, provide opportunities to practice these skills in session. During role plays, participants monitor stigmatizing beliefs that may interfere with communication or pursuing goals.
  Interventions: Behavioral: Self-stigma intervention

INTERVENTIONS:
Behavioral: Self-stigma intervention — Be Outspoken and Overcome Stigmatizing Thoughts (BOOST) is a group-based intervention integrating cognitive behavioural therapy (CBT) and peer support to reduce or prevent the internalization of stigma in early psychosis. The BOOST group will last for 4 weeks and consists of two 1-hour sessions per week. Participants will be assessed prior to the first group, following the final group, six months after the group ends, and twelve months after the group ends.
  Other Names: Be Outspoken and Overcome Stigmatizing Thoughts (BOOST)

SUMMARY:
Internalized stigma, (i.e. the application of negative stereotypes about a diagnostic group to one's self) is a strong predictor of recovery and quality of life for individuals with psychosis. Be Outspoken and Overcome Stigmatizing Thoughts (BOOST) is an evidence-based intervention aimed at improving internalized stigma, self-esteem, and quality of life for those with psychosis. The proposed research expands BOOST's program by adding additional therapeutic methods and material, and adopting the use of virtual care methods to: (a) increase the generalization of treatment effects, (b) examine long-term treatment effects, and (C) provide rural Ontario communities with remote treatment access.

DETAILED DESCRIPTION:
Internalized stigma, defined as the application of negative stereotypes about a diagnostic group to one's self, is a strong predictor of quality of life and recovery in schizophrenia and other psychoses, accounting for over half the variance. However, few effective interventions for self-stigma have been developed and even fewer individuals have access to these services.

Be Outspoken and Overcome Stigmatizing Thoughts (BOOST) is an evidence-based intervention developed by the research team that has significantly improved internalized stigma, self-esteem, and quality of life for young people with psychosis. This group therapy was co-created and is co-facilitated by people with lived experience with psychosis specifically for the early psychosis population. The proposed research expands this intervention by examining the efficacy of group delivery through virtual methods that could allow us to reach individuals that are unlikely to attend regular in-person sessions for a variety of reasons.

Psychotic disorders are among the most highly stigmatized mental health conditions. Over 50% of individuals with schizophrenia and other psychoses report significant internalization of these stigmatizing attitudes. Internalized stigma is defined as the application of societally held stereotypes about the illness to one's self. It is associated with a broad array of significant psychosocial consequences including reduced social functioning, isolation, and reduced rates of recovery. Internalized stigma is also associated with serious decrements in self-esteem, self-efficacy, and hope. Reducing internalized stigma has been recognized as such a critical factor in recovery from psychosis that both the World Health Organization and National Institute for Health and Care Excellence prioritize the reduction of stigma to improve recovery from psychosis.

Despite the clear importance of reducing internalized stigma in psychosis, few interventions have been developed to reduce internalized stigma about mental illness. Only a single intervention had previously been developed to specifically reduce internalized stigma among individuals in the early stages of psychosis. None of these internalized stigma interventions have demonstrated strong evidence for efficacy. The current approaches to reducing internalized stigma have focused almost exclusively on psychoeducation about psychosis, without evidence-based therapeutic techniques, and with treatment later in illness, when self-stigma has already set in. The investigators developed Be Outspoken and Overcome Stigmatizing Thoughts (BOOST), a group-based intervention integrating cognitive behavioural therapy (CBT) and peer support to reduce or prevent the internalization of stigma in early psychosis. Peer support is an especially important intervention for psychosis as peer support workers provide personal examples to normalize experiences that clients are having. Peer support has been demonstrated to improve social functioning and recovery for individuals with psychosis. Thus, the investigators propose that the combination of these approaches would be ideal to reduce internalized stigma.

In the initial pilot study[13], BOOST demonstrated significant improvements in internalized stigma, self-esteem, and quality of life. Despite BOOST demonstrating the largest effect size improvement on internalized stigma of any intervention currently evaluated (Cohen's d = 0.76), this was a small non-randomized sample, so the investigators would like to build the evidence base for the intervention and examine the breadth of treatment effects.

Proposed Solution Description:

BOOST is an 8-session group intervention, delivered over 4 weeks, near the time of psychosis onset. BOOST is the only intervention that integrates cognitive behavioural therapy with peer support, and these two intervention work synergistically to reduce internalized stigma. Interactive sessions are co-led by a psychologist or doctoral level psychology student and a peer support worker with lived experience. Sessions 1-4 focus on dispelling stigmatizing myths about psychosis and evaluating the accuracy of group members or societies stigmatizing beliefs in order to normalize experiences associated with and reactions to the symptoms of psychosis. Exercises include identifying the effects of self-labelling, evaluating self-stigmatizing beliefs, and testing the dimensionality of experiences associated with psychosis. All of these exercises are designed to help participants develop new ways of thinking that more accurately reflect the evidence, to build confidence in their capacity to recognize and modify negative self-attributions, and provide hope for the future. Sessions 5-8 teach behavioural approaches for self-empowerment through social skills training, development of assertiveness skills, and goal setting. Discussions in group are focused on the verbal and non-verbal characteristics of passive, aggressive, and assertive communication, as well as how to develop social communication and problem-solving skills. Role-plays that are specific to young people with psychosis, which were co-developed with people with lived experience, provide opportunities to practice these skills in session. During role plays, participants monitor stigmatizing beliefs that may interfere with communication or pursuing goals. Throughout each session, the peer support worker uses both prepared and spontaneous examples from their experiences of internalized stigma, negative beliefs, communication, and recovery in order to normalize experiences and instill hope. This is an interactive intervention designed for individuals of all cultural backgrounds. Although the internalized stigma belief content may be different in different cultures, the process of evaluating and normalizing experiences is consistent across demographic and geographic factors. Inclusion of a wide geographic sample in this project enhances the ability to generate a diverse set of content during group discussions.

Preliminary BOOST findings show large statistical effects in changing variables predictive of future suicidal ideation and behaviour, such as self-esteem and internalized stigma. The goal of the proposed research is to conduct a trial to examine how effective this group treatment for self-stigma, co-developed and co-facilitated by service users is when delivered through virtual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder or any other psychotic disorder
* Must be 18-35 years of age
* Know how to use a computer and telephone
* Not abusing drugs or alcohol
* Can read and speak English

Exclusion Criteria:

* Individuals enrolled in a cognitive behavioural therapy program in the last 6 months
* Individuals with neurological disease or neurological damage
* Individuals with medical illnesses that can change neurocognitive function
* Individuals with a medical history of a head injury with loss of consciousness
* Physical handicaps that would prevent an individual from engaging in the BOOST program

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Internalized stigma | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  This project will assess how virtual BOOST treatment changes psychological factors associated with recovery. The primary outcome measure is internalized stigma as measured by the Internalized Stigma of Mental Illness Scale.

SECONDARY OUTCOMES:
Self-Injurious Thoughts and Behaviours Interview Self-Report | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Cognition associated with risk of suicide
Interpersonal Hopelessness Scale | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Cognition associated with hopelessness
Interpersonal Needs Questionnaire | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Interpersonal needs measure
Rosenberg Self-Esteem Scale | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Self-esteem measure
Patient Health Questionnaire | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Depression symptom severity measure
Psychache Scale | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Depression symptom severity measure
Generalized Anxiety Disorder scale (GAD-7) | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Self-reported anxiety measure
Satisfaction with Life Scale | Participants will be assessed at baseline, and assessed for changes immediately following the treatment and at 6 months and 12 months post treatment.
  Quality of life measure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Bowie, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No